CLINICAL TRIAL: NCT04093791
Title: MAMA NO STRESS Project. The Effects of the "HAPPY MAMA" Intervention: a Field Randomized Trial
Brief Title: MAMA NO STRESS Project. The Effects of the "HAPPY MAMA" Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuseppe La Torre, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 80209930587
Record Dates: First submitted 2019-06-11; First posted 2019-09-18 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Depression, Postpartum; Stress, Psychological; Postpartum Sadness; Self Efficacy; Mother-Infant Relations
Keywords: postpartum; stress; depression; self efficacy; Mother-Infant Relations
MeSH Terms: conditions — Depression, Postpartum; Stress, Psychological; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided in three groups: the one that will follow the collective intervention (G); the one that will follow the Individual Intervention (I) and the control group, that will receive no intervention (C)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Collective Intervention "G" (Experimental): HAPPY MAMA intervention will follow the following steps: listening and establishing relationship phases; analysis of the problems; definition of the problem and the goal of intervention.
  The duration will be of 3.5 hours in one day and the intervention will happen in "Sapienza" University of Rome, in a group of 15 women.
  This group fill in an on line questtionarie for four times, the first before the intervention.
  Interventions: Behavioral: Collective Intervention "G"
- Individual Intervention "I" (Experimental): The same intervention of "G" group (HAPPY MAMA), but at individual level and the intervention will happen at the participants' house.
  This group fill in an on line questtionarie for four times, the first before the intervention.
  Interventions: Behavioral: Individual Intervention "I"
- Control group "C" (No Intervention): The women from this group will not receive any intervention. This group fill in an on-line questtionarie for four times.

INTERVENTIONS:
Behavioral: Collective Intervention "G" — The steps are:
  1. Listening/establishing relationship. This step is characterized by listening and understanding the critical points from the new mothers. The operator maintains a nonjudgmental approach encouraging the women to describe the need for behavioral change.
  2. Analysis. The situation must be carefully evaluated, considering the discomfort and emotional distress. The stress situation will be described in a subjective way and they will assign a grade of discomfort for each problem.
  3. Assessment. The operator will carry out a multidimensional evaluation of the mothers within the dyad. The operator will evaluate the strategies implemented by the mothers to face problems and the reasons of the failures.
  4. Summary and goal of the intervention. The problems detected by the operator will be explained and summarized to the participants. The operator explores ways to implement change.
  Other Names: HAPPY MAMA G intervention
  Arms: Collective Intervention "G"
Behavioral: Individual Intervention "I" — The steps are:
  1. Listening/establishing relationship. This step is characterized by listening and understanding the critical points from the new mother. The operator maintains a nonjudgmental approach encouraging the woman to describe the need for behavioral change.
  2. Analysis. The situation have be carefully evaluated, considering the discomfort and emotional distress. The stress situation will be described in a subjective way, and she will assign a grade of discomfort for each problem.
  3. Assessment. The operator will carry out a multidimensional evaluation of the mothers within the dyad. The operator will evaluate the strategies implemented by the mother to face problems and the reasons of the failures.
  4. Summary and goal of the intervention. The problems detected by the operator will be explained and summarized to the participants. The operator explores ways to implement change.
  Other Names: HAPPY MAMA I intervention
  Arms: Individual Intervention "I"

SUMMARY:
This study evaluates the effects of a postpartum intervention in increasing the maternal well-being and self-efficacy of Italian women in the first one to six months after childbirth, as well as in reducing postpartum depression and stress.

The intervention will use the motivational interviewing against high levels of daily stress. One third of participants will be exposed to a 3,5 hours group intervention approximately 1 month after delivery, one third will be exposed to an individual intervention in the same period and one third will receive no intervention. Participants will be followed with stress and depression questionnaires.

DETAILED DESCRIPTION:
Aim

The aim of this study is to assess the effectiveness of an intervention, called "HAPPY MAMA", in reducing postpartum stress level, increasing the parenting self-efficacy and the maternal well-being of Italian women in the first one to six months after childbirth.

Design of the study

The study will be an experimental pilot field trial. The present research will be a multi-centric study to be conducted in three different hospitals in Rome. The CONSORT statement will be followed to perform the research.

Eligibility criteria for participants

The following eligibility criteria will be applied:

* Participant must be a woman aged 18 years old or older;
* Participant must be able to communicate in Italian.

They following exclusion criteria will be applied:

* women will be excluded from the study if they or their babies have serious health problems;
* the baby was born at <37 weeks gestation, weighed <2500 g;
* the baby has the APGAR score <7 immediately after birth. Participants will be recruited from the Obstetrics Units of the following Hospitals: Teaching Hospital Umberto 1, Teaching Hospital "Casilino" and "S. Giovanni Calibita Fatebenefratelli".

Furthermore for organizational reasons, only mothers that live in Rome will be enrolled.

The hospital recruitment of participants will be conducted at 0 to 3 days postpartum by the researchers and research nurses using a brochure explaining the aim of the study.

The recruitment period will in two weeks. Prior to study participation all women who agree to participate will be asked to sign a written consent form and to provide a contact phone number and email.

Randomization

After taking the consent, the participants will be divided into three groups:

* group that will follow the "Collective intervention group," that will be called "G";
* group that will follow the "Individual intervention group," that will be called "I";
* control group that will be called "Control group" (C).

The allocation of the women in the groups will be randomly. The investigators will create a random number sequence using Epicalc 2000. A researcher will assign the participants to the groups following the number sequence as described below:

* Multiples of three (3,6,9,12, etc.) in G;
* Multiples of three+1 (1, 4, 7,10, etc.) in I;
* Multiple of three+2 (2, 5, 8, 11, etc.)in C.

The groups will be matched for followed variables:

* age (>31 years, 31 is the mean age of Italian women at childbirth (ISTAT, 2017));
* vaginal delivery (Yes/No).

Data collection

The recruitment period will be of two weeks. During the delivery hospital (T0), the researchers will ask to sign consent forms from each participant and they will collect the demographics information for matching and performing the randomization.

During T0 phase an unique code will be assigned to each women (for example a keyword composed using the first three letter of her name and the last four numbers of her telephone number). A check will be done of the uniqueness, and in case of overlap an adjustment it will be done.

For organizational reasons, one researcher has a paper sheet that reported the codes associated to the women's names.

After the recruitment and the randomization phase, a message that contains the link to the questionnaire will be sent by phone.

The questionnaire is created using a Google form.

The questionnaire will be administered four times:

* At T1: About 30 days weeks after the hospital delivery and 15 days, the last women recruited:

  * For G: the questionnaire will be administered on-line with a phone message with a link to the questionnaire. The message will be sent 2/3 days before the collective intervention. The meeting will be performed about15 days after the last women recruited;
  * For I: the questionnaire will be administered on-line with a phone message with a link to the questionnaire. The message will be sent 2/3 days before the individual intervention. The single intervention will be performed 30 days after the hospital delivery (the 30 days is a hypothesis made considering that in the G group means the time that has elapsed since of giving birth to the intervention is the median range between 2 or 4 weeks).
  * For women in the C group, the questionnaire will be administered online with a phone message with a link to the questionnaire. The message will be sent 30 days after the delivery.
* At T2: About two months after delivery:

  * For G: the questionnaire will be administered online with a phone message with a link to the questionnaire. The message will be sent about one month after the collective intervention;
  * For I: the questionnaire will be administered online with a phone message with a link to the questionnaire. The message will be sent one month after the individual intervention;
  * For C: the questionnaire will be administered online with a phone message with a link to the questionnaire. The message will be sent two months after the delivery.
* At T3: the questionnaire will be administered online with a phone message with a link to the questionnaire. The message will be sent three months after the delivery (T3);
* At T4: the questionnaire will be administered online with a phone message with a link to the questionnaire. The message will be sent six months after the delivery.

Questionnaire

The online questionnaire will be used to obtain socio-demographic data, characteristics of breastfeeding practice, mother's confidence about their ability to successfully raise children, and the information on stress and depression.

In order to find the measurements of stress level, self-efficacy and depression in the mothers, a literature search on Pubmed using following search terms "maternal stress, depression, self-efficacy AND (questionnaire or index or inventory)" was conducted on 25th March 2019.

The search display 53 papers, after an analysis of the abstract and the full text the researchers have composed a questionnaire that includes the following three validated scales:

* the Karitane Parenting Confidence Scale (KPCS) as a measure of the perceived parental self-efficacy (PPSE), defined as ''beliefs or judgments a parent holds of their capabilities to organize and execute a set of tasks related to parenting a child''. The 15-item scale, grounded in self-efficacy theory, was developed to assess PPSE of parents with infants aged 0-12 months. Factor analysis revealed a three-factor structure, composed of efficacy, support, and child development. An Italian version of the questionnaire will be used.
* the Parental Stress Scale (PSS). The PSS scale consisted of 18 items rated on a 5-point Likert scale. The total score was obtained by summing up the value for each item. A higher score indicates a higher level of parental stress. An Italian version of the questionnaire will be used.
* the Italian version of the Edinburgh Postnatal Depression Scale (EPDS). This questionnaire is used to measure maternal depressive symptoms. The EPDS is a self-report screening measure to detect symptoms of postpartum depression. Scores >12 on the EPDS are correlated with a diagnosis of major depressive disorder (MDD).

At the baseline, the questionnaire includes additionally a section of demographic variables. The following characteristics will be collected: age, civil status (single or not), employment (student/ worker/ no worker), educational level (middle school/ high school/ university), the birth date, primipara (yes/ no), number of children living at home and age, vaginal birth (yes/no), Italian Region where she lives, city where she lives, ethnicity.

The women will be interviewed four times, always by phone call:

For G and I groups: About 2/3 weeks after the last women recruited and 2/3 days before the intervention (T1); about two month after the delivery that it is about one month after the intervetion(T2); three months after the delivery (T3); six months after the delivery (T4).

For the C group: About 2/3 weeks after the delivery(T1); about 30 days after delivery(T2); three months after the delivery (T3); six months after the delivery (T4).

HAPPY MAMA Intervention

Collective level (G)

The training carried out by a childcare worker and midwives with high experience in childcare and home interventions, includes educational and mindfulness training and simulations of typical events. Given the importance of communication skills training and better outcomes in studies where skills practice has taken place, the interventionists developed their skills through patient simulation and role-play scenarios with one another and the facilitators before interacting with study participants.

The phases of the intervention can be educational and support-based, as needed. The educational phase aims to provide information, demonstrations, and discussions.

1. Objectives The objective of the HAPPY MAMA intervention is to explore the effects of early proactive parenting support strategies on mothers' confidence, stress, and mood. The ultimate goal is to share and increase awareness of one's abilities: control and autonomy are important for the final step of the process, the last step wants to put new mothers in a position to implement strategies, and be able to pursue goals to restore mental well-being
2. Structure

The phases of the intervention can be educational and support-based, as needed. The educational phase aims to provide information, demonstrations, and discussions while supporting phase aimed at providing social support, counseling, or consultation. The intervention follows several steps:

1. Listening and establishing relationship phases. The first step is characterized by listening and understanding the critical points from the new mother.

   This requires the use of listening skills, empathy, authenticity, and acceptance. The operator maintains a nonjudgmental approach and allows the woman to determine the need for behavioral change, rather than offering unsolicited advice on the need for change.
2. Analysis of the problems The situation must be carefully evaluated, considering the discomfort and emotional distress. The stress situation will be described in a subjective way, from the new mother/s, and she/they will assign a grade of discomfort for each problem.
3. Assessment. The operator will carry out a multidimensional evaluation of the mother/s within the dyad. The operator will evaluate the strategies implemented by the new mother/s to face problems and the reasons of their failures; for example: how she routinely handles organizational problems, how she experiences breastfeeding if there is a lack of sleep and how she considers her family and support network.

   The evaluation will have to consider the environment as a whole, with attention to facilitators and barriers.
4. Definition of the problem and the goal of the intervention The problems detected by the operator will be explained and summarized to the participant/s. The operator only explores ways to implement change once the woman/women expresses the desire and confidence to change.

The shared identification of the mother/s' priority will lead to the definition of a tailored plan aimed at achieving specific goals such as the reduction of the stress levels, the decline of the sleep deprivation (hours of sleep per night), optimization of breastfeeding (number, duration and quality), increased well-being (mental health, physical health).

Strategies of concrete action and planned behavior will be provided adapted to the context and styles of women/woman's coping.

Time Length of the intervention will be 3 hours in one day.

Location and number of partecipans Group interventions will take place at the Department of Public Health and Infectious Diseases of "Sapienza" University of Rome. Number of participants: 20 (max).

Individual interventions will be carried out at the women's home.

Descriptive statistics will be performed using frequencies and percentage for qualitative variables. Moreover the measures of central tendency (mean or median) and of variability (Standard Deviation, SD, interquartile range, IQR) will be computed in order to describe the quantitative variables in each groups.

The univariate analysis will be used to compare groups (G, I and C) versus primary and secondary outcomes. In particular, Kruskall Wallis's test will be applied to assess possible difference of stress scores between the three groups; Chi-square's test will be applied to assess possible independence between the three groups versus categorical variables, too.

The tests for paired samples will be used to assess the possible changes of the stress score during the follow-up of the G and I groups (baseline, T1, versus 2(T2), 3 (T3) and 6 (T4)months after the intervention).

A linear regression model will be used in order to assess possible significant predictors of the outcomes and a R2 will be computed as the indicator of the goodness of fit of the model.

The significant level is fit at p<0.05.

ELIGIBILITY:
The following eligibility criteria will be applied:

* Participant must be a woman aged 18 years old or older;
* Participant must be able to communicate in Italian.

They following exclusion criteria will be applied:

* women will be excluded from the study if they or their babies have serious health problems;
* the baby was born at <37 weeks gestation, weighed <2500 g;
* the baby has the APGAR score <7 immediately after birth (17).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Assessing a change of the Parental Stress Scale (PSS): The main outcome measures are the Parental Stress Scale (PSS) for change between the baseline and the follow-up (four time points). | 4 weeks after the delivery or 2/3 days before the intervention; 2 months after delivery or 2 weeks after the intervention; 3 months after delivery; 6ths after delivery.
  The PSS scale consisted of 18 items rated on a 5-point Likert scale. The total score was obtained by summing up the value for each item. A higher score indicates a higher level of parental stress. An Italian version of the questionnaire will be used.
  A follow-up of the PSS score will be computed.

SECONDARY OUTCOMES:
Assessing a change of the Karitane Parenting Confidence Scale (KPCS). The secondary outcome measures are theKaritane Parenting Confidence Scale (KPCS) for change between the baseline and the follow-up (four time points). | 4 weeks after delivery or 2/3 days before the intervention; 2 months after delivery or 2 weeks after the intervention; 3 months after delivery; 6 months after delivery.
  a measure of the perceived parental self-efficacy (PPSE), defined as ''beliefs or judgments a parent holds of their capabilities to organize and execute a set of tasks related to parenting a child''. The 15-item scale, grounded in self-efficacy theory (20), was developed to assess PPSE of parents with infants aged 0-12 months. Factor analysis revealed a three-factor structure, composed of efficacy, support, and child development. An Italian version of the questionnaire will be used.
  A follow-up of the PSS score will be computed.
Assessing a change of the Edinburgh Postnatal Depression Scale (EPDS). The secondary outcome measures are the Edinburgh Postnatal Depression Scale (EPDS) for change between the baseline and the follow-up (four time points). | 4 weeks after delivery or 2/3 days before the intervention; 2 months after delivery or 2 weeks after the intervention; 3 months after delivery; 6 months after delivery.
  10 screening questions, answered by the mother on telephone interview, that can indicate whether a parent has symptoms that are common with depression and anxiety. Score goes from 0-30, being 30 the most severe postnatal depression symptoms.
  A follow-up of the PSS score will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Mannocci, Principal Investigator — University "La Sapienza", Department of Public Health and Infectious Diseases

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] APGAR V. A proposal for a new method of evaluation of the newborn infant. Curr Res Anesth Analg. 1953 Jul-Aug;32(4):260-7. No abstract available. PMID 13083014
- [Background] Bennett AE, Kearney JM. Factors Associated with Maternal Wellbeing at Four Months Post-Partum in Ireland. Nutrients. 2018 May 14;10(5):609. doi: 10.3390/nu10050609. PMID 29757937
- [Background] Beresford BA. Resources and strategies: how parents cope with the care of a disabled child. J Child Psychol Psychiatry. 1994 Jan;35(1):171-209. doi: 10.1111/j.1469-7610.1994.tb01136.x. PMID 8163627
- [Background] Carpiniello B, Pariante CM, Serri F, Costa G, Carta MG. Validation of the Edinburgh Postnatal Depression Scale in Italy. J Psychosom Obstet Gynaecol. 1997 Dec;18(4):280-5. doi: 10.3109/01674829709080700. PMID 9443138
- [Background] Cheng CY, Li Q. Integrative review of research on general health status and prevalence of common physical health conditions of women after childbirth. Womens Health Issues. 2008 Jul-Aug;18(4):267-80. doi: 10.1016/j.whi.2008.02.004. Epub 2008 May 12. PMID 18468922
- [Background] Cheng CY, Fowles ER, Walker LO. Continuing education module: postpartum maternal health care in the United States: a critical review. J Perinat Educ. 2006 Summer;15(3):34-42. doi: 10.1624/105812406X119002. PMID 17541458
- [Background] Coates R, Ayers S, de Visser R. Women's experiences of postnatal distress: a qualitative study. BMC Pregnancy Childbirth. 2014 Oct 14;14:359. doi: 10.1186/1471-2393-14-359. PMID 25315742
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Gallagher L, Begley C, Clarke M. Determinants of breastfeeding initiation in Ireland. Ir J Med Sci. 2016 Aug;185(3):663-668. doi: 10.1007/s11845-015-1333-2. Epub 2015 Jul 15. PMID 26174153
- [Background] Kahn RS, Zuckerman B, Bauchner H, Homer CJ, Wise PH. Women's health after pregnancy and child outcomes at age 3 years: a prospective cohort study. Am J Public Health. 2002 Aug;92(8):1312-8. doi: 10.2105/ajph.92.8.1312. PMID 12144990
- [Background] Kristensen IH, Simonsen M, Trillingsgaard T, Pontoppidan M, Kronborg H. First-time mothers' confidence mood and stress in the first months postpartum. A cohort study. Sex Reprod Healthc. 2018 Oct;17:43-49. doi: 10.1016/j.srhc.2018.06.003. Epub 2018 Jun 25. PMID 30193719
- [Background] O'Hara MW, McCabe JE. Postpartum depression: current status and future directions. Annu Rev Clin Psychol. 2013;9:379-407. doi: 10.1146/annurev-clinpsy-050212-185612. Epub 2013 Feb 1. PMID 23394227
- [Background] Perez-Blasco J, Viguer P, Rodrigo MF. Effects of a mindfulness-based intervention on psychological distress, well-being, and maternal self-efficacy in breast-feeding mothers: results of a pilot study. Arch Womens Ment Health. 2013 Jun;16(3):227-36. doi: 10.1007/s00737-013-0337-z. Epub 2013 Mar 20. PMID 23512648
- [Background] Coates R, de Visser R, Ayers S. Not identifying with postnatal depression: a qualitative study of women's postnatal symptoms of distress and need for support. J Psychosom Obstet Gynaecol. 2015;36(3):114-21. doi: 10.3109/0167482X.2015.1059418. Epub 2015 Jul 1. PMID 26135567
- [Background] Tarkka MT, Paunonen M, Laippala P. Factors related to successful breast feeding by first-time mothers when the child is 3 months old. J Adv Nurs. 1999 Jan;29(1):113-8. doi: 10.1046/j.1365-2648.1999.00868.x. PMID 10064289
- [Background] Wagnild GM, Young HM. Development and psychometric evaluation of the Resilience Scale. J Nurs Meas. 1993 Winter;1(2):165-78. PMID 7850498
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Benvenuti P, Ferrara M, Niccolai C, Valoriani V, Cox JL. The Edinburgh Postnatal Depression Scale: validation for an Italian sample. J Affect Disord. 1999 May;53(2):137-41. doi: 10.1016/s0165-0327(98)00102-5. PMID 10360408